CLINICAL TRIAL: NCT04743752
Title: Obstructive Sleep Apnea Influences Efficacy of Anti-Programmed-Death-1-Based Immunotherapy Against Non-Small Cell Lung Cancer - A Prospective Observational Cohort Study
Brief Title: Obstructive Sleep Apnea Influences Efficacy of PD-1-Based Immunotherapy Against Non-Small Cell Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Jing MA, Prof.&MD, Peking University First Hospital
Other Study IDs: 2020-405
Record Dates: First submitted 2021-01-30; First posted 2021-02-08 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Obstructive Sleep Apnea; Non-small Cell Lung Cancer
MeSH Terms: conditions — Sleep Apnea, Obstructive; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fecal and peripheral blood specimens
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group OSA+NSCLC: According to the baseline sleep monitor results, participants will be divided into Group OSA+NSCLC if apnea hypopnea index(AHI) no less than 15.
- Group NSCLC: According to the baseline sleep monitor results, participants will be divided into Group NSCLC if apnea hypopnea index(AHI) less than 15.

SUMMARY:
This prospective, observational cohort study aims to explore the influence of obstructive sleep apnea(OSA) on the efficacy of PD-1-based immunotherapy in patients with non-small cell lung cancer(NSCLC). Patients who had no prior treatment for advanced NSCLC and are intended to receive PD-1/PD-L1 antibody will be recruited. According to sleep monitor results, participants will be divided into Group NSCLC and Group OSA+NSCLC. Primary outcome is the objective remission rate(ORR).

DETAILED DESCRIPTION:
This is a single-center, prospective, observational cohort study. Patients who had no prior treatment for advanced NSCLC and are intended to receive PD-1/PD-L1 antibody will be recruited and followed for 4 years. According to the baseline sleep monitor results, participants will be divided into Group NSCLC(AHI<15), and Group OSA+NSCLC(AHI≥15), and then explore the influence of obstructive sleep apnea on the efficacy of PD-1-based immunotherapy. The baseline level of white blood cell count (WBC); absolute neutrophil count (ANC); absolute lymphocyte count (ALC); ANC to ALC (ANC:ALC) ratio; interleukin 6 (IL-6); C-reactive Protein (CRP) in peripheral blood, lymphocytes classification and count by flow cytometry, and gut microbiome analysis by quantitative metagenomics will also be measured to further search for the possible mechanisms. Primary outcome is the objective remission rate (ORR), secondary outcomes include overall survival (OS) and progression free survival (PFS).

The study protocol has been approved by the Peking University First Hospital Institutional Review Board (IRB). Any protocol modifications will be submitted for the IRB review and approval.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed, advanced NSCLC
2. Participants with no prior treatment for advanced NSCLC
3. Measurable disease as defined by RECIST v1.1
4. Eligible to receive first-line treatment including PD-1 antibody
5. Adequate hematologic and end organ function

Exclusion Criteria:

1. Severe infection within 4 weeks prior to recruitment.
2. Significant organ dysfunction or other serious diseases.
3. Previous or current OSA related treatment, including oral appliance, surgery, mechanical ventilation therapy.
4. Illness or condition that interferes with the participant's capacity to understand, follow and/or comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had no prior treatment for advanced NSCLC and are intended to receive PD-1/PD-L1 antibody will be recruited and followed for 4 years.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | From date of randomization until the date of first documented progression, assessed up to 48 months
  ORR, the percentage of complete response (CR) or partial response (PR) according to RECIST 1.1 standard definition.CR: disappearance of all target and non-target lesions and (if applicable) normalization of tumor marker level; or reduction in short axis of any pathological lymph nodes (whether target or non-target) to less than (<) 10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters; or persistence of one or more non-target lesion(s) and/or (if applicable) maintenance of tumor marker level above the normal limits.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  PFS was defined as the time from recruitment to the first occurrence of progressive disease(PD) or death due to any cause. PD: at least a 20 percent increase in the sum of diameters of target lesions, taking as reference the smallest sum on study, including baseline, and an absolute increase of at least 5 mm; appearance of one or more new target or non-target lesions; or unequivocal progression of existing non-target lesions.
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 48 months
  OS was defined as the time from the date of enrollment to the date of death due to any cause.
Compared the baseline sleep monitor results between Group NSCLC and Group OSA+NSCLC. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Record baseline AHI, oxygen desaturation index (ODI), lowest saturation by pulse oximetry (SpO2)<90%, obstructive apnea index (OAI), central apnea index(CAI), the longest apnea duration, then compare between Group NSCLC and Group OSA+NSCLC.
Factors associated with ORR in NSCLC patients | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Cox regression analysis will be used to identify predictors of ORR.
Factors associated with OS and PFS in NSCLC patients | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Univariate and multivariate Cox proportional hazards models will be used to identify predictors of PFS and OS.
Compared the baseline level of lymphocytes classification and count between Group NSCLC and Group OSA+NSCLC. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Record baseline lymphocytes classification and count in peripheral blood, then compare between Group NSCLC and Group OSA+NSCLC.
Compared the baseline level of inflammatory biomarkers between Group NSCLC and Group OSA+NSCLC. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Record baseline interleukin 6 (IL-6) and C-reactive Protein (CRP) in peripheral blood, then compare between Group NSCLC and Group OSA+NSCLC.
The association between OSA and baseline inflammatory biomarkers, peripheral lymphocytes classification and count. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  The Spearman correlation test will be used to identify the association between sleep monitor results and the baseline inflammatory biomarkers, peripheral lymphocytes classification and count, including AHI, ODI, lowest SpO2, SpO2<90%, OAI, CAI, the longest apnea duration
Compared the baseline gut microbiome between Group NSCLC and Group OSA+NSCLC. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  Record baseline gut microbiome by metagenomic shotgun sequencing, then compare between Group NSCLC and Group OSA+NSCLC.
The association between OSA and the diversity of gut microbiome. | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  The Spearman correlation test will be used to identify the association between sleep monitor results and the diversity of gut microbiome, including AHI, ODI, lowest SpO2, SpO2<90%, OAI, CAI, the longest apnea duration.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ma, MD, Study Chair — Peking University First Hospital; Guangfa Wang, MD, Study Director — Peking University First Hospital; Yuan Cheng, Study Director — Peking University First Hospital; Ligong Nie, Study Director — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No